CLINICAL TRIAL: NCT06871371
Title: The Comparison of the Effects of Low and Medium Flow Anesthesia on Haemodynamics, Arrhytmia Risk and Cerebral Oxygenation in Laparoscopic Cholecystomy Cases
Brief Title: Low and Moderete Flow Anaesthesia on Haemodynamics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Senay Goksu, specialist, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: LFATUGCE
Record Dates: First submitted 2025-01-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemodynamics Instability; Arrhythmias Cardiac; Cerebral Oxygenation
Keywords: Low-Medium Flow Anesthesia, Hemodynamics, Oxygenation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- low flow anesthesia (Active Comparator): Maintenance of anaesthesia with low-flow anaesthesia
  Interventions: Device: Sevoflurane (Volatile Anesthetic); Device: low- medium flow anesthetic machine
- Medium Flow Anesthesia (Active Comparator): Maintenance of anaesthesia with medium-flow anaesthesia
  Interventions: Device: Sevoflurane (Volatile Anesthetic); Device: low- medium flow anesthetic machine

INTERVENTIONS:
Device: Sevoflurane (Volatile Anesthetic) — Both groups will be given sevoflurane and one group will be given low current anesthesia and the other group will be given medium flow anesthesia.
Device: low- medium flow anesthetic machine — The study aims to compare the effects of low and normal flow sevoflurane anesthesia on the frontal QRS-T angle and cerebral oxygenation in laparoscopic cholecystectomy surgery.

SUMMARY:
The study topic investigates the potential advantages of low-flow anesthesia in terms of physiological protection and resource saving.

DETAILED DESCRIPTION:
The study aims to compare the effects of low and normal flow sevoflurane anesthesia on the frontal QRS-T angle and cerebral oxygenation in laparoscopic cholecystectomy surgery. The primary objective was to evaluate the effects of low-flow anesthesia on hemodynamic stability and arrhythmia risk; the secondary objective was to compare the total sevoflurane consumption in both methods.

ELIGIBILITY:
Inclusion Criteria:

* being ASA1-2 status
* between the ages of 18-70
* who are planned for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients who refuse to give informed consent
* Pregnant and breastfeeding patients
* Morbidly obese patients (Body mass index over 40)
* Patients with uncontrolled diabetes mellitus, with serious cardiovascular, pulmonary, renal, hepatic disease, obstructive sleep apnea, with electrolyte imbalance- Those with a history of alcohol or drug abuse, with perioperative hemodynamic instability
* Patients using drugs known to prolong myocardial repolarization
* inability to increase SPO2 above 95 despite necessary intervention

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
the effects of low-flow anesthesia on hemodynamic stability | in 2 months
  The primary objective was to detect the adverse effects of low-flow anesthesia on hemodynamic stability and arrhythmia risk

SECONDARY OUTCOMES:
the cerebral oxygenation | in 2 months
  The primary objective was to detect the adverse effects of low-flow anesthesia on cerebral oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: SENAY GOKSU, MD, Principal Investigator — UMRANIYE E R HOSPITAL
Locations (1):
- Umraniye Education and research hospital, Istanbul, Turkey (Türkiye)